CLINICAL TRIAL: NCT05274971
Title: Dietary Management and Aerobic Exercise on 24-hour Ambulatory Blood Pressure in Subjects with Prehypertension and Drug-naïve Stage 1 Hypertension: Randomized, Single-blinded Clinical Trial
Brief Title: Diet and Exercise on Ambulatory Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: The Korean Vascular Research Working Group (Unknown)
Responsible Party: Principal Investigator, Soon Jun Hong, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Daphne
Record Dates: First submitted 2022-02-05; First posted 2022-03-11 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-04

CONDITIONS: Prehypertension
Keywords: Prehypertension; aerobic exercise; Dietary management
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Intervention Model Description: Experimental group versus Control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active management group (Experimental): Active dietary management and aerobic exercise training. Subjects will receive assessment and education of DASH diet (0, 4, and 8 weeks), with active aerobic exercise training (1 hour everyday exercise, at least 5 times per week for 12 weeks) (aerobic exercise education at baseline, 4, and 8 weeks after randomization). Each set of aerobic exercise consists of 10 minutes warm-up, 40 minutes moderate-intensity treadmill trotting, and 10 minutes cooldown. Telephone counseling at 2, 6, and 10 weeks after randomization.
  Interventions: Other: Active dietary management and aerobic exercise training.
- Control group (No Intervention): Subjects will not receive education and recommendation of dietary management and aerobic exercise training.

INTERVENTIONS:
Other: Active dietary management and aerobic exercise training. — Active dietary management and aerobic exercise training.
  Arms: Active management group

SUMMARY:
This is a multicenter, randomized, single-blinded clinical trial investigating the effect of dietary management and active aerobic exercise training on reduction of 24-hour ambulatory blood pressure in subjects with prehypertension and drug-naïve stage 1 hypertension.

DETAILED DESCRIPTION:
Most guidelines recommend lifestyle modifications such as exercise or dietary programs for stage 1 hypertension or prehypertension, before initiation of antihypertensive drug treatment. Epidemiological and observational studies have shown that cardiovascular risk increases progressively from blood pressure levels as low as 115/75 mmHg and that patients with prehypertension or stage 1 hypertension are likely to progress to hypertension requiring medications. From a previous clinical trial, a 12-week aerobic exercise program reduced 24-hour and daytime ambulatory blood pressure in patients with resistant hypertension. Aerobic exercise and DASH (Dietary Approaches to Stop Hypertension) diet are currently recommended in subjects with prehypertension and stage 1 hypertension without a clear randomized, controlled clinical trial. The present trial, thus, seeks to evaluate the effect of dietary management and active aerobic exercise training, preferably moderate-intensity exercise, on 24-hour ambulatory blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Prehypertension or grade 1 hypertension, defined as a systolic blood pressure of 130 to 159 mm Hg and/or a diastolic blood pressure of 85 to 99 mm Hg
* Patients without previous use of anti-hypertensive medication

Exclusion Criteria:

* Patients under anti-hypertensive medications
* Patients with suspected or confirmed secondary hypertension
* Patients with abnormal liver function tests (transaminases more than three times the upper limit of normal)
* Patients without aerobic exercise tolerance
* Patients under hormone replacement therapy or other steroids
* Patients with peripheral edemas and/or baseline serum creatinine level above 2.0 mg/dL
* Patients with medical conditions that potentially affect blood pressure, including neurological disorders, gastrointestinal diseases, or malignancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour ambulatory systolic blood pressure | from baseline to 12 weeks
  Change in 24-hour ambulatory systolic blood pressure
Change in 24-hour ambulatory diastolic blood pressure | from baseline to 12 weeks
  Change in 24-hour ambulatory diastolic blood pressure
Change in daytime ambulatory systolic and diastolic blood pressure | from baseline to 12 weeks
  Change in daytime ambulatory systolic and diastolic blood pressure
Change in nighttime ambulatory systolic and diastolic blood pressure | from baseline to 12 weeks
  Change in nighttime ambulatory systolic and diastolic blood pressure
Change in office systolic and diastolic blood pressure | from baseline to 12 weeks
  Change in office systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Change in arterial stiffness | from baseline to 12 weeks
  augmentation index
Change in arterial stiffness | from baseline to 12 weeks
  pulse wave velocity
Change in serum renin level | from baseline to 12 weeks
  Change in serum renin level
Change in serum angiotensin converting enzyme (ACE) level | from baseline to 12 weeks
  Change in serum angiotensin converting enzyme (ACE) level
Change in circulating endothelial and inflammatory biomarkers | from baseline to 12 weeks
  interleukin-6
Change in circulating endothelial and inflammatory biomarkers | from baseline to 12 weeks
  interleukin-18
Change in circulating endothelial and inflammatory biomarkers | from baseline to 12 weeks
  Tumour Necrosis Factor alpha
Change in circulating endothelial and inflammatory biomarkers | from baseline to 12 weeks
  high sensitivity-C-reactive protein
Change in circulating endothelial and inflammatory biomarkers | from baseline to 12 weeks
  Soluble Vascular Cell Adhesion Molecule-1 (sVCAM-1)
Change in circulating endothelial and inflammatory biomarkers | from baseline to 12 weeks
  Soluble intercellular adhesion molecule-1 (sICAM-1)
Change in circulating endothelial and inflammatory biomarkers | from baseline to 12 weeks
  Plasminogen activator inhibitor-1

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Chul Sung, Study Chair — Kangbuk Samsung Hospital, Sungkyunkwan University School of Medicine, Seoul, South Korea
Locations (1):
- Korea University Anam Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lim S, Hong SJ, Kim JH, Cha JJ, Joo HJ, Park JH, Yu CW, Lim DS, Shin JH, Lee JY, Lim YH, Kim SH, Sung KC. Dietary management and aerobic exercise counselling on blood pressure control in subjects with prehypertension and drug-naive stage 1 hypertension: a randomized clinical trial. Sci Rep. 2025 Dec 29;15(1):45683. doi: 10.1038/s41598-025-20828-7. PMID 41462029